CLINICAL TRIAL: NCT04302441
Title: A Study to Evaluate Vinorelbine Plus Capecitabine Combined With Trastuzumab as the Adjuvant Treatment of HER2 Positive Patients Following Neoadjuvant Chemotherapy
Brief Title: A Study to Evaluate Vinorelbine Plus Capecitabine Combined With Trastuzumab for HER2 Positive Patients Following Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-162-9
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: non-pCR; HER2 positive; vinorelbine; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NXH group (Experimental): Patients should receive four cycles of NXH regimen (vinorelbine at 25 mg/m2 iv infusion on day 1 and day 8 plus capecitabine 1000mg/m2, po, bid, d1-d14, 21 days per cycle, trastuzumab at 6mg/kg iv infusion on day1 every 3 weeks to 1 year).
  Interventions: Drug: Vinorelbine; Drug: Capecitabine
- H group (No Intervention): Patients should receive trastuzumab at 6mg/kg iv infusion on day1 every 3 weeks to 1 year.

INTERVENTIONS:
Drug: Vinorelbine — vinorelbine 25mg/m2 on day 1 and 8,every 3 weeks
  Arms: NXH group
Drug: Capecitabine — Capecitabine 1000mg/m2, po, bid, d1-d14, 21 days per cycle
  Arms: NXH group

SUMMARY:
This study aims to evaluate vinorelbine plus capecitabine combined with trastuzumab versus trastuzumab alone as the adjuvant Treatment of HER2 positive patients following neoadjuvant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Patients with histologically confirmed unilateral invasive ductal carcinoma(according to WHO histologically type)
* Tumor clinical staged as IIB-IIIB before neoadjuvant chemotherapy (according to the 7th AJCC edition).
* After standard treatment (at least 6 cycles) of neoadjuvant chemotherapy (plan formulated by the attending doctor, including anthracycline and paclitaxel drugs combined with trastuzumab), assessed by the surgery, the original site for non - pCR (MP class 1-4) or lymph nodes are still positive for patients.
* No gross or microscopic tumor residual after resection.
* Patients with Her2 receptor positive (Specific definition: immunohistochemical detection of Her2 3+ or Her2 2 + but after FISH or CISH tested is positive).
* No evidence of distant metastasis in the clinical or radiological aspects of preoperative. examination,that is M0.
* Patients without peripheral neuropathy or I peripheral neurotoxicity.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
* Patients recovered well after surgery, at least 1 weeks after the operation.
* Adequate marrow: White blood cells count≥3000/μL,neutrophil count ≥1500/μL, hemoglobin ≥9g/dL and platelet count ≥75000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ 1.5ULN.
* Adequate renal function: Serum creatinine ≤ 1.5ULN.
* Contraception during the treatment of child-bearing women.
* Adequate cardiac function :Left ventricular ejection fraction (LVEF) > 50%.
* Patients must be informed of the investigational nature of this study and give written informed consent.
* Patients without serious heart, lung, liver, kidney and other important organs disease history.
* Patients have good compliance.

Exclusion Criteria:

* Patients with bilateral breast cancer or carcinoma in situ(DCIS/LCIS).
* Metastasis of any part except axillary lymph nodes.
* Clinical or imaging suspicion of the contralateral breast is malignant but not confirmed, requiring biopsy.
* There have been malignant tumors (except for basal cell carcinoma and carcinoma in situ of cervix) in the last five years, including breast cancer.
* Patients have been enrolled in other clinical trials.
* Patients with severe systemic illnesses and/or uncontrolled infections are unable to join the study.
* Patients with severe cardio-cerebrovascular disorders (e.g., unstable angina pectoris, chronic heart failure, uncontrollable hypertension >160/100mmgh, myocardial infarction or cerebrovascular accident) in the first 6 months of randomization.
* Pregnant lactating women (child-bearing women must be negative for pregnancy test within 14 days prior to first delivery, if positive, the pregnancy should be excluded by ultrasound.)
* Child-bearing women who are unwilling to take effective contraceptive measures in the course of research.
* Patients with mental illness, cognitive impairment, inability to understand test protocols and side effects, and those who fail to complete the trial programme and follow-up work (a systematic assessment is required before the trial).
* Persons without personal freedom and independent civil capacity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 550 (Estimated)
Dates: Start 2016-11-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 year
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer

SECONDARY OUTCOMES:
Recurrence free survival | 3 year
  Recurrence free survival is calculated from surgery to the first recurrence
Distant disease free survival | 3 year
  Distant disease free survival is calculated from surgery to the first distant metastasis.
Overall survival | 5=3 year
  Overall survival is calculated from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No